CLINICAL TRIAL: NCT06534463
Title: The Effectiveness and Safety of Different Treatment Modalities in Real-World Clinical Practice Among Chinese Patients with Marginal Zone Lymphoma: a Prospective, Observational, Multi-center Study
Brief Title: Registry Study of Chinese Patients with Marginal Zone Lymphoma (MOTIVE)
Acronym: MOTIVE
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Deputy director of hospital, Ruijin Hospital
Other Study IDs: MOTIVE
Record Dates: First submitted 2024-07-21; First posted 2024-08-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Cohort: Including newly diagnosed marginal zone lymphoma (MZL) and relapse/refractory MZL participants who meet the treatment indications for MZL and are about to undergo MZL treatment.
  Interventions: Other: All treatment regimen selections and usage will be determined by the physician based on clinical practice and/or the respective drug labels in China.

INTERVENTIONS:
Other: All treatment regimen selections and usage will be determined by the physician based on clinical practice and/or the respective drug labels in China. — The dosage and duration of any drug in this study will be determined by the physician based on local clinical practice and local drug labels. The drugs in this study include, but are not limited to, Obinutuzumab, Rituximab, Bruton tyrosine kinase inhibitors, and Lenalidomide. In this non-interventional study, all treatment drug usage will be determined by the physician based on clinical practice and/or the respective drug labels in China.

SUMMARY:
This study aims to evaluate real-world treatment modalities and their corresponding effectiveness and safety in Chinese patients with marginal zone lymphoma, while also exploratively analyzing patient characteristics and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as MZL
* Meet the treatment indications for MZL

Exclusion Criteria:

* Any reason that, in the investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are about to undergo marginal zone lymphoma(MZL) treatment (i.e., those who have been recommended for and intend to receive MZL treatment at the time of signing the informed consent form)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to approximately 60 months)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Response Rate | End of treatment visit (approximately 6 months)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Complete Response Rate | End of treatment visit (approximately 6 months)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Time to Next Treatment | From the start of treatment to the initiation of next-line treatment (up to approximately 60 months)
  From the start of treatment to the initiation of next-line treatment
Duration of Response | Baseline up to data cut-off (up to approximately 60 months)
  Time from first occurrence of documented complete response or partial response to disease progression/relapse, or death from any cause for participants, whichever occurs first.
Duration of Complete Response | Baseline up to data cut-off (up to approximately 60 months)
  Time from the first occurrence of a documented complete response to the date of progression, relapse, or death from any cause, whichever occurs first.
Overall survival | Baseline up to data cut-off (up to approximately 60 months)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to data cut-off (up to approximately 60 months)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

OTHER OUTCOMES:
Health-Related Quality of Life assessed with EORTC QLQ-C30 questionaire | Baseline up to data cut-off (up to approximately 60 months)
  Patient-reported outcomes using The European Organization for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30) .
Health-Related Quality of Life assessed with EORTC QLQ-NHL-LG20 questionaire | Baseline up to data cut-off (up to approximately 60 months)
  Patient-reported outcomes using The European Organization for Research and Treatment of Cancer Quality of Life questionnaire including 20 items for patients with low-grade non-Hodgkin lymphoma (EORTC QLQ-NHL-LG20).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No